CLINICAL TRIAL: NCT00473785
Title: Community Outreach Heart Health and Risk Reduction Trial
Brief Title: CVD Risk Reduction Trial
Acronym: COHRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSFO4857; HSFO Grant # 4857
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular disease; Prevention; Lifestyle
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Group-based motivational interviewing
Behavioral: Individual CVD-risk factor feedback
Behavioral: Education for protective health behavior change

SUMMARY:
The purpose of this study is to provide lifestyle counselling for protective health behavior (exercise, diet, smoking cessation) to small groups (6-8 subjects) via teleconference. The sample includes individuals at elevated risk for cardiovascular disease (CVD) as well as individuals with established CVD. Our hypothesis is that telephone-based lifestyle counselling will (1) significantly increase protective lifestyle behavior (diet, exercise, smoke-free living) and (2) significantly reduce CVD risk factors at 6-month follow-up.

DETAILED DESCRIPTION:
COHRT was a 2 parallel-group randomized controlled trial that was designed to assess the efficacy of a community outreach strategy for cardiovascular disease (CVD) risk reduction among individuals at elevated risk for CV events. Randomization was stratified for diagnosis of CHD, type 1 or 2 diabetes, sex, and clinical depression, and blocked within our northern, rural, and urban recruitment sites. A 2X3 mixed factorial design was utilized: 2 Groups (Usual Care, UC/Lifestyle Counselling,LC) X 3 Intervals (Baseline, post-treatment, 6-month follow-up). All subjects received personal CVD risk factor feedback and standardized handouts on heart healthy lifestyle change. The LC group received 6 weekly 1-hour sessions of lifestyle counseling that was provided via teleconference in small groups (4-8 persons). Group facilitators were trained in a manualized protocol of motivational interviewing that was designed for CVD risk reduction through lifestyle change. Weekly supervision was also provided. We hypothesized that the LC group (vs. UC) would significantly increase protective health behavior (exercise, diet, smoke-free living) at post-treatment and 6-month follow-up. The secondary hypothesis was that LC would significantly reduce (1) CVD risk factors, (SBP, DBP, total cholesterol, LDL cholesterol), (2) 10-year absolute risk among subjects without CVD, and (3) significantly increase quality of life as measured by symptoms of depression, psychological stress, and social support.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 74 years of age,
* Diagnosis of CVD or Type 1 or 2 diabetes, or
* ≥2 of the following CVD risk factors:

  * Confirmed diagnosis of hypertension,
  * Dyslipidemia,
  * Males aged ≥55 years/females aged ≥60 years,
  * Family history of CHD or stroke;
  * Current smoker, or
  * BMI ≥ 27.

Exclusion Criteria:

* Diagnosis of clinically significant cardiac complications (e.g. arrhythmia, unstable angina) or a congenital cardiac condition;
* Major psychiatric illness (e.g. psychosis), history of alcohol or drug dependence within the previous year, or residence in a non-private setting.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 827 (Actual)
Dates: Start 2002-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Psychometric assessment of change in exercise, diet and smoking | Post-treatment and 6-month follow-up

SECONDARY OUTCOMES:
SBP, DBP, total cholesterol, HDL, LDL, triglycerides and 10-year absolute CVD risk | 6-month follow-up
Psychometric assessment of symptoms of depression, psychological stress, and social support. | post-treatment and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Nolan, PhD, Principal Investigator — University Health Network/University of Toronto
Locations (3):
- Canada (3):
  - Laurentian University / Sudbury and District Health Unit, Greater Sudbury, Ontario
  - Grey-Bruce Health Unit, Owen Sound, Ontario
  - University Health Network / Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Grace SL, Barry-Bianchi S, Stewart DE, Rukholm E, Nolan RP. Physical activity behavior, motivational readiness and self-efficacy among Ontarians with cardiovascular disease and diabetes. J Behav Med. 2007 Feb;30(1):21-9. doi: 10.1007/s10865-006-9080-5. Epub 2006 Nov 16. PMID 17109217